CLINICAL TRIAL: NCT03798808
Title: The Impact of an Innovative Family and Web-based Nutrition Intervention to Increase Vegetable, Fruit, and Dairy Intakes in Children With Overweight or Obesity: A Single-blinded Randomized Family Clustered Intervention
Brief Title: Family and Web-based Nutrition Intervention to Increase Vegetable, Fruit, and Dairy Intakes in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Vicky Drapeau, Professor, Laval University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NUTRIATHLON-2015-259 R-2
Record Dates: First submitted 2019-01-08; First posted 2019-01-10 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Diet Habit
Keywords: vegetables, fruits, dairy, children, habits
MeSH Terms: conditions — Feeding Behavior; Habits | interventions — Fruit; Vegetables; Dairy Products

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family Nutriathlon group (Experimental): Web-based nutrition program (encouraging consumption of fruits, vegetables and dairy products through an online platform)
  Interventions: Other: Consumption of fruits, vegetables and dairy products
- Control group (No Intervention): General nutrition guidelines (e.g. following Canada's Food Guide)

INTERVENTIONS:
Other: Consumption of fruits, vegetables and dairy products — Family Nutriathlon was an eight-week, family-based nutrition program where children and their parents were encouraged to reach individual and team goals with respect to the quantity and variety of fruit, vegetable and dairy product consumption.
  Arms: Family Nutriathlon group

SUMMARY:
Considering the high prevalence of childhood obesity worldwide, effective interventions are needed . Parental involvement in interventions and the use of web-based modalities appear to be promising approaches. The aim of the study was to evaluate the efficacy of an innovative family and Web-based nutrition intervention called "Family Nutriathlon" on consumption of vegetables and fruit and dairy products and/or alternatives and on diet quality among children and their parents.

DETAILED DESCRIPTION:
Forty-three families, with at least one child with a BMI >85th percentile, participated in either the intervention (n=24) or control group (n=19) over an 8-week period. Families in the intervention (Family Nutriathlon) will participated in a nutrition challenge that aimed to increase their consumption and variety of fruits and vegetables and dairy products by recording their daily intakes using a Web-based platform. Families in the control group received recommendations based on general nutrition guidelines. Three follow-ups with a dietitian once every two weeks via Skype to assess progress were scheduled. A three-day food record was completed at baseline (week 0), immediately after (week 8) and 6 months after the intervention. A two-way repeated measures analysis of variance was used to assess changes in consumption of fruits and vegetables and dairy products, diet quality and dietary intakes between groups and over time.

ELIGIBILITY:
All inclusion/exclusion criterion were the same between the two projects (including the intervention) except for the inclusion of a child living with obesity or overweight.

Children were aged between 8 and 16 years, but there was no age limit for parents.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Dietary intakes and diet quality | 8 weeks
  Fruit, vegetable and dairy product consumption and diet quality as measured by the Nutrient-Rich Foods Index

SECONDARY OUTCOMES:
Anthropometric measurements | Weeks 0, 9 and 18-36 (follow-up)
  Body weight, height and body mass index

REFERENCES:
- [Derived] Drapeau V, Harvey AA, Jacob R, Provencher V, Panahi S. The impact of a family web-based nutrition intervention to increase fruit, vegetable, and dairy intakes: a single-blinded randomized family clustered intervention. Nutr J. 2022 Dec 20;21(1):75. doi: 10.1186/s12937-022-00825-6. PMID 36539753